CLINICAL TRIAL: NCT02993900
Title: A Clinical Trial To Evaluate Image-Guided Gynecologic Brachytherapy In The MR Simulator Suite
Brief Title: Image-Guided Gynecologic Brachytherapy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: J1660; IRB00098525 (Other: JHM IRB); R21CA167800 (NIH)
Record Dates: First submitted 2016-11-30; First posted 2016-12-15 (Estimated); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Cervical Cancer; Uterine Cancer; Vaginal Cancer; Vulvar Cancer; Bladder Cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms; Uterine Neoplasms; Vaginal Neoplasms; Vulvar Neoplasms; Urinary Bladder Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Image-Guided Brachytherapy (Experimental): Magnetic Resonance Imaging (MRI) guided brachytherapy Procedure: Image-Guided Brachytherapy
  Interventions: Device: Image-Guided Brachytherapy

INTERVENTIONS:
Device: Image-Guided Brachytherapy — Brachytherapy will be precisely inserted with the assistance of magnetic resonance (MRI) scans

SUMMARY:
This research is being done to evaluate multimodality imaging, including magnetic resonance imaging-guided therapy (MRT), as a possible treatment for gynecologic cancers. The therapy takes place in the Department of Radiation Oncology at the Johns Hopkins SKCCC. The purpose of this study is to investigate the ability of MRI to successfully guide the placement of the brachytherapy applicator necessary to treat participants' gynecologic cancer. The Investigators want to see if the use of MRI will do a better job of assessing the tumor at the time of brachytherapy than the routinely used CT scan. The Investigators also want to determine if the use of MRI will enable doctors to reduce the radiation dose received by the body during the process of treating the tumor.

DETAILED DESCRIPTION:
The goal of this trial is to assess how magnetic resonance imaging (MRI) may be used to improve tumor and normal tissue volume delineation, reducing toxicity and recurrence in gynecologic brachytherapy. The Investigators will compare dosimetric values to the organs at risk (OAR) with CT versus MRI planning. The Investigators anticipate that MR-planned cases will have lower OAR doses than standard CT-based cases due to more conformal planning. The Investigators will determine dose thresholds for radiation-related toxicity after treatment. The Investigators will compare toxicity rates at 6 months, 1 and 2 years after treatment, thereby enabling improved recommendations on dose limits to the OAR.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have histologically or cytologically confirmed carcinoma. Central pathology review is not required; however, pathology will be reviewed at the SKCCC at Johns Hopkins.
* Site/Stage
* Any patient eligible for internal implantation without MR guidance will be considered eligible for this protocol. Standard criteria for internal implantation include:
* Carcinoma of the cervix: Stage I-IVA or vaginal recurrence
* Carcinoma of the uterus: Stage IIIB (vaginal involvement), inoperable, or vaginal recurrence
* Carcinoma of the vagina: Stage I-IVA or vaginal recurrence
* Carcinoma of the vulva: Stage I-IVA or recurrence
* Carcinoma of the urethra based on treating physician's discretion
* Patients who have received prior radiation or chemotherapy may be enrolled on this study.
* Age > 18 years. Children do not develop these malignancies and therefore are not considered candidates for this trial.
* Life expectancy of greater than 6 months.
* ECOG performance status of <2 or greater, based on treating physician's discretion
* MRI of the pelvis or PET-CT within 4 months before registration
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Absolute neutrophil count < 500 at the time of enrollment
* A history of metal in the head or eyes

Ages: 18 Years to 100 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2016-12-15 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Dosing changes | 3 years
  To quantify the relative reduction of dose to rectum, sigmoid and bladder obtained after MR Simulator Suite-guided placement, as compared to standard CT guided treatment based on historical information and literature review.

SECONDARY OUTCOMES:
The rate of treatment-related toxicity | 3 months, 6 months and 1 year
  To determine the rate of treatment-related toxicity within 3 months, 6 months and 1 year after MR Simulator Suite-guided placement.
Time to local failure | 1 year and 2 year
  To determine the local failure rates at 1 year and 2 year after MR Simulator Suite-guided placement.
Rate of survival | 1 year and 2 year
  To determine the overall survival rates at 1 year and 2 year after MR Simulator Suite-guided placement.

CONTACTS AND LOCATIONS:
Overall Officials: Akila Viswanathan, M.D., Principal Investigator — Johns Hopkins Department of Radiation Oncology
Locations (1):
- The SKCCC at Johns Hopkins, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No